CLINICAL TRIAL: NCT01679899
Title: Effect of Anti-diabetic Drugs on Bone Metabolism and Glycemic Variability.A Comparison Between Vildagliptin and Gliclazide MR
Brief Title: Effect of Anti-diabetic Drugs on Bone Metabolism and Glycemic Variability
Acronym: BoneGlyc
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centro de Diabetes Curitiba Ltda (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BoneGlyc
Record Dates: First submitted 2012-09-02; First posted 2012-09-06 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Type 2 Diabetes Mellitus; Menopause; Osteoporosis; Osteopenia
Keywords: diabetes; type 2 diabetes mellitus; osteopenia; osteoporosis; glycemic variability; bone markers; osteocalcin; NTX; CTX; BALP
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Osteoporosis; Bone Diseases, Metabolic; Diabetes Mellitus | interventions — Vildagliptin; Gliclazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vildagliptin (Experimental): Vildagliptin 50 mg bid for 12 months
  Interventions: Drug: Vildagliptin
- Gliclazide MR (Active Comparator): Gliclazide MR 60 or 120mg once a day for 12 months
  Interventions: Drug: Gliclazide MR

INTERVENTIONS:
Drug: Vildagliptin — Vildagliptin 50mg bid orally for 12 months
  Other Names: Galvus
  Arms: Vildagliptin
Drug: Gliclazide MR — Gliclazide MR 60 or 120mg orally for 12 months
  Other Names: Diamicron MR
  Arms: Gliclazide MR

SUMMARY:
This is a Monocentric, Prospective, Randomized, Open-label, Comparative, Phase IV Study, to compare the effects of Vildagliptin and Gliclazide MR on Markers of Bone Remodeling, Bone Mineral Density and Glycemic Variability in Postmenopausal Women with Type 2 Diabetes.

A total of 38 women with documented Type 2 Diabetes and menopause will be enrolled. The active treatment will include a 50 mg dose of vildagliptin OD twice a day. As comparator, gliclazide MR will be administered at a dose of 60 to 120 mg OD once a day.

DETAILED DESCRIPTION:
This is a Monocentric, Prospective, Randomized, Open-label, Comparative, Phase IV Study, to compare the effects of Vildagliptin and Gliclazide MR on Markers of Bone Remodeling, Bone Mineral Density and Glycemic Variability in Postmenopausal Women with Type 2 Diabetes.

Target population of clinical trial subjects A total of 38 women with documented Type 2 Diabetes and menopause will be enrolled. To be as close to a real life scenario as possible, clinical trial subjects which are treated with glucose-lowering medication (except incretin or sulfonylurea based therapies) and treatment-naive subjects will be included.

Investigational Product, posology and method of administration The active treatment will include a 50 mg dose of vildagliptin OD twice a day.

Comparator, posology and method of administration As comparator, gliclazide MR will be administered at a dose of 60 to 120 mg OD once a day.

Treatment duration The study will have an expected total duration of 18 months, 12 months of active treatment.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent form obtained before any study-related activity. Study-related activities are any procedure that would not be performed during the normal treatment of the patient.
* All study subjects must be women diagnosed with type 2 diabetes based on current guidelines of Sociedade Brasileira de Diabetes (SBD - Brazilian Society of Diabetes) and/or American Society of Diabetes (ADA) and they should have all the following criteria:

  * Age ≥ 40 years old.
  * HbA1c ≥ 6.5% at randomization.
* Menopause defined as:
* Absence of menstruation for at least 12 months in patients with an intact uterus, or
* FSH level greater than 30 mIU/mL in a hysterectomized patient and/or,
* FSH level greater than 30 mIU/mL in a patient with surgical menopause.

Exclusion Criteria:

* Acute vascular event (cardiac, cerebral or peripheral) for at least 2 months of randomization.
* Patient on chronic dialysis and/or renal transplantation and/or serum creatinine > 1.5 mg/dL.
* Patients with HIV, severe autoimmune disease or chronic treatment with oral steroids (> 30 consecutive days).
* Current or previous treatment (within 6 months) with incretin (DPP-IV inhibitor or GLP-1 analog) within 6 months prior to randomization.
* Current or previous treatment with pioglitazone or rosiglitazone within 12 months prior to randomization.
* Sustained arterial hypertension > 180/100 mm Hg.
* Body mass index (BMI) > 50 kg/m².
* HbA1c ≥ 9,5% at randomization.
* Transaminases (AST (SGOT) and ALT (SGPT)) > 2.5 x upper limit of normal.
* Chronic liver disease or alcoholic liver disease.
* LDL-cholesterol > 250 mg/dL (> 6.48 mmol/L).
* Triglycerides > 1000 mg/dL (> 11.3 mmol/L).
* HDL-cholesterol < 25 mg/dL (< 0.64 mmol/L).
* Levels of 25-OH-vitamin D < 20ng/mL at randomization
* Abnormal levels of PTH, cortisol, IGF-1 or GH at randomization
* Prescription of any investigational medication within one year before the screening visit (visit 1), unless there is a direct benefit to the study subject, at the discretion of the investigator.
* History of previous fracture
* Pregnant or breastfeeding patients.
* Previous participation on this study.
* Individuals at risk for poor adherence to the protocol or medication.
* Any condition that makes the patient unable to complete the study within 12 months.

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Markers of bone remodeling | 6 months
  Primary outcome is to compare the effect of vildagliptin with gliclazide MR on markers of bone remodeling. The outcome variables are the blood levels of:
  1. Osteocalcin (OC)
  2. Bone-specific alkaline phosphatase (BALP)
  3. Carboxy-terminal telopeptide of type I collagen (CTX)
  4. Amino-terminal telopeptide of type I collagen (NTX)

SECONDARY OUTCOMES:
Bone mineral density of lumbar spine and femur by X-ray absorptiometry | 12 months
  To compare the effect of vildagliptin with gliclazide MR on bone mineral density of lumbar spine and femur by X-ray absorptiometry after 12-month treatment.
Glycemic variability | 6 months
  To compare the effect of vildagliptin with gliclazide MR on glycemic variability measured by MAGE method (mean amplitude of glycemic excursion) using a continuous glucose monitoring system
Calcitonin | 12 months
  Dosage of serum calcitonin

OTHER OUTCOMES:
Levels of aminotransferases | 6 months
  Dosage of alanine aminotransferase (ALT, SGOT) and aspartate aminotransferase (AST, SGPT)

CONTACTS AND LOCATIONS:
Overall Officials: Andre GD Vianna, MD, Study Chair — Centro de Diabetes Curitiba
Locations (1):
- Centro de Diabetes Curitiba, Curitiba, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vianna AGD, de Lacerda CS, Pechmann LM, Polesel MG, Marino EC, Borba VZC, Barreto FC. Vildagliptin has the same safety profile as a sulfonylurea on bone metabolism and bone mineral density in post-menopausal women with type 2 diabetes: a randomized controlled trial. Diabetol Metab Syndr. 2017 May 15;9:35. doi: 10.1186/s13098-017-0232-2. eCollection 2017. PMID 28515791